CLINICAL TRIAL: NCT00554788
Title: A Trial of Intensive Multi-Modality Therapy for Extra-Ocular Retinoblastoma
Brief Title: Combination Chemotherapy, Autologous Stem Cell Transplant, and/or Radiation Therapy in Treating Young Patients With Extraocular Retinoblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARET0321; NCI-2009-00421 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARET0321; CDR0000573987; COG-ARET0321; ARET0321 (Other: Children's Oncology Group); ARET0321 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Extraocular Retinoblastoma
MeSH Terms: interventions — Bone Marrow Transplantation; Stem Cell Transplantation; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Radiotherapy; Radiation; Thiotepa; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, radiotherapy, autologous SCI) (Experimental): INDUCTION: Patients receive vincristine IV; cisplatin IV; cyclophosphamide IV; and G-CSF SC beginning on day 3 and continuing until blood counts recover.
  CONSOLIDATION (stage 4a or 4b disease only): Patients receive carboplatin IV; thiotepa IV; and etoposide IV.
  AUTOLOGOUS STEM CELL INFUSION (stage 4a or 4b disease only): Patients undergo autologous stem cell infusion on day 0 and receive G-CSF SC beginning on day 1 and continuing until blood counts recover.
  RADIOTHERAPY: Patients with stage 2 or 3 disease (orbital and/or regional involvement) undergo radiotherapy to sites that were initially involved beginning within 42 days after the start of course 4 of induction chemotherapy. Patients with stage 4a or 4b disease undergo radiotherapy to sites initially involved based on response beginning approximately 42 days after autologous stem cell infusion.
  Interventions: Procedure: Autologous Bone Marrow Transplantation; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carboplatin; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Etoposide; Biological: Filgrastim; Procedure: In Vitro-Treated Peripheral Blood Stem Cell Transplantation; Radiation: Radiation Therapy; Drug: Thiotepa; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Autologous Bone Marrow Transplantation — Undergo peripheral blood stem cell or bone marrow transplant
  Other Names: ABMT; Autologous Blood and Marrow Transplantation; Autologous Bone Marrow Transplant; Autologous Marrow Transplantation
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo peripheral blood stem cell or bone marrow transplant
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Biological: Filgrastim — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Procedure: In Vitro-Treated Peripheral Blood Stem Cell Transplantation — Undergo peripheral blood stem cell or bone marrow transplant
  Other Names: in vitro-treated PBPC transplantation; in vitro-treated peripheral blood progenitor cell transplantation
Radiation: Radiation Therapy — Undergo radiotherapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Thiotepa — Given IV
  Other Names: 1,1',1''-Phosphinothioylidynetrisaziridine; Girostan; N,N', N''-Triethylenethiophosphoramide; Oncotiotepa; SH 105; SH-105; SH105; STEPA; Tepadina; Tepylute; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase III trial is studying the side effects and how well giving combination chemotherapy together with autologous stem cell transplant and/or radiation therapy works in treating young patients with extraocular retinoblastoma. Giving chemotherapy before an autologous stem cell transplant stops the growth of tumor cells by stopping them from dividing or killing them. After treatment, stem cells are collected from the patient's blood and/or bone marrow and stored. More chemotherapy is given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy. Radiation therapy uses high energy x-rays to kill tumor cells. Giving radiation therapy after combination chemotherapy and/or autologous stem cell transplant may kill any remaining tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To estimate the proportion of 3 groups of patients with extraocular retinoblastoma (stage 2 and 3: regional extra-ocular disease;, stage 4a: disseminated metastatic disease not involving the central nervous system [CNS]; or stage 4b: patients with CNS disease) who achieve long-term event-free survival after treatment with aggressive multimodality therapy compared to historical controls.

II. To estimate the response rate to the induction phase of the regimen. III. To evaluate the toxicities associated with this regimen.

OUTLINE:

INDUCTION CHEMOTHERAPY: Patients receive vincristine intravenously (IV) on days 0, 7, and 14, cisplatin IV over 6 hours on day 0, cyclophosphamide IV over 1 hour and etoposide IV over 1 hour on days 1 and 2, and filgrastim (G-CSF) subcutaneously (SC) beginning on day 3 and continuing until blood counts recover.

Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of induction chemotherapy, patients with stage 2 or 3 disease who have at least a partial response proceed to radiotherapy. Patients with stage 4a or 4b disease who have at least a partial response proceed to high-dose consolidation chemotherapy and autologous stem cell infusion.

STEM CELL HARVESTING (stage 4a or 4b disease only): Peripheral blood stem cells (preferred) or bone marrow cells are collected after at least 1 course of induction chemotherapy.

HIGH-DOSE CONSOLIDATION CHEMOTHERAPY (stage 4a or 4b disease only): Patients receive carboplatin IV over 4 hours on days -8 to -6 and thiotepa IV over 3 hours and etoposide IV over 3 hours on days -5 to -3.

AUTOLOGOUS STEM CELL INFUSION (stage 4a or 4b disease only): Patients undergo autologous stem cell infusion on day 0. Patients then receive filgrastim subcutaneously (SC) beginning on day 1 and continuing until blood counts recover.

RADIOTHERAPY: Patients with stage 2 or 3 disease (orbital and/or regional involvement) undergo radiotherapy to sites that were initially involved beginning within 42 days after the start of course 4 of induction chemotherapy. Patients with stage 4a or 4b disease undergo radiotherapy to sites initially involved based on response beginning approximately 42 days after autologous stem cell infusion. Patients with stage 4a disease who achieve a complete response to induction chemotherapy or with less than 5 mm of residual tumor at the time of planned irradiation, or patients with stage 4b disease who achieve a complete response to induction chemotherapy do not undergo radiotherapy.

After completion of study therapy, patients are followed every 3 months for 1 year and then annually thereafter for 9 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic or cytologic verification of extra-ocular retinoblastoma; extra-ocular disease includes orbital disease, optic nerve involvement at the surgical margin, regional nodal disease, and/or overt distant metastatic disease (at sites such as bone, bone marrow, liver and/or the central nervous system); patients with trilateral retinoblastoma will also be included in this protocol

  * Patients with a CNS lesion consistent with trilateral or stage 4b disease may be enrolled without tissue confirmation if (1) unequivocal leptomeningeal disease is present on brain or spine magnetic resonance imaging (MRI) scan and/or (2) the primary tumor is at least 2 cm in diameter, predominantly solid, and demonstrates enhancement on the post-gadolinium images; however, even in such cases surgery should be given serious consideration
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* No prior chemotherapy or radiotherapy for the extra-ocular retinoblastoma may have been administered prior to entering this study; prior treatment (chemotherapy and/or radiation therapy) for intra-ocular retinoblastoma is permissible
* Peripheral absolute neutrophil count (ANC) >= 750/uL

  * If the ANC and/or platelet count are not adequate, but due to bone marrow metastatic disease, these criteria will be waived
* Platelet count >= 75,000/uL (transfusion independent)

  * If the ANC and/or platelet count are not adequate, but due to bone marrow metastatic disease, these criteria will be waived
* Creatinine clearance OR radioisotope glomerular filtration rate >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 0.4 mg/dL (1 month to < 6 months of age)
  * 0.5 mg/dL (6 months to < 1 year of age)
  * 0.6 mg/dL (1 years to < 2 years of age)
  * 0.8 mg/dL (2 years to < 6 years of age)
  * 1.0 mg/dL (6 years to < 10 years of age)
  * 1.2 mg/dL (10 years to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 years to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (>= 16 years of age)
* Total bilirubin =< 1.5 times upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 x upper limit of normal (ULN)
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) for human studies must be met

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2008-05-06 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira J Dunkel, Principal Investigator — Children's Oncology Group
Locations (73):
- United States (66):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Morristown Medical Center, Morristown, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Hospital de Pediatria Juan P Garrahan, Buenos Aires, Argentina
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Instituto De Oncologia Pediatrica, São Paulo, Brazil
- Canada (2):
  - IWK Health Centre, Halifax, Nova Scotia
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- Children's Cancer Hospital, El Saida Zenab, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Dunkel IJ, Piao J, Chantada GL, Banerjee A, Abouelnaga S, Buchsbaum JC, Merchant TE, Granger MM, Jubran RF, Weinstein JL, Saguilig L, Abramson DH, Krailo MD, Rodriguez-Galindo C, Chintagumpala MM. Intensive Multimodality Therapy for Extraocular Retinoblastoma: A Children's Oncology Group Trial (ARET0321). J Clin Oncol. 2022 Nov 20;40(33):3839-3847. doi: 10.1200/JCO.21.02337. Epub 2022 Jul 12. PMID 35820112

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 2/3 Patients: Patients with orbital disease (including microscopic trans-scleral invasion seen on enucleation pathology), optic nerve margin (+), and/or regional nodal disease, but no other sites of metastases. Stage 2 and 3 patients will receive Induction chemotherapy and External Beam Radiation Therapy, but will not receive Consolidation therapy (High-Dose Chemotherapy with Stem Cell Rescue).
- Stage 4a Patients: Patients with overt distant metastatic disease (such as bone, bone marrow, and/or liver) but no detectable CNS involvement. Patients will receive Induction chemotherapy, Stem Cell Harvesting, Consolidation with Stem Cell Rescue, and depending on response to Induction chemotherapy, possibly External Beam Radiation Therapy.
- Stage 4b Patients: Patients with overt CNS involvement (brain parenchyma, leptomeninges and CSF cytology). Patients with trilateral retinoblastoma will be included. Patients will receive Induction chemotherapy, Stem Cell Harvesting, Consolidation with Stem Cell Rescue, and depending on response to Induction chemotherapy, possibly External Beam Radiation Therapy.
Period: Overall Study
Arm/Group | Stage 2/3 Patients | Stage 4a Patients | Stage 4b Patients
Started | 21 | 18 | 21
Completed | 14 | 12 | 7
Not Completed | 7 | 6 | 14
Not completed — Adverse Event | 0 | 1 | 2
Not completed — Lost to Follow-up | 4 | 3 | 3
Not completed — Physician Decision | 1 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Refusal of further protocol therapy | 0 | 1 | 1
Not completed — Progressive disease | 0 | 0 | 3
Not completed — Ineligible | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 2/3 Patients | Stage 4a Patients | Stage 4b Patients | Total
Number analyzed (Participants) | 21 | 18 | 21 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.24 (1.36) | 3.96 (2.27) | 2.91 (1.83) | 3.34 (1.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 14 | 27
  Male | 17 | 9 | 7 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 8 | 23
  Not Hispanic or Latino | 13 | 10 | 13 | 36
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 5 | 10
  White | 11 | 11 | 12 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 4 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 14 | 13 | 41
  Canada | 1 | 0 | 0 | 1
  Argentina | 3 | 4 | 2 | 9
  Egypt | 3 | 0 | 4 | 7
  Brazil | 0 | 0 | 1 | 1
  Chile | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: The probability of surviving patients who did not experience events at 1 year following enrollment. An event is defined as relapse, second malignancy, or death from any cause.
Time Frame: At 1 year
Population: Ineligible patients were excluded from analysis
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Stage 2/3 Patients | Stage 4a Patients | Stage 4b Patients
Number analyzed (Participants) | 19 | 18 | 20
Probability | 88 [60 to 97] | 83 [55 to 94] | 28 [10 to 49]

2. Secondary Outcome: Response Rate to the Induction Phase of the Regimen
Description: This study used a modified version of the international criteria for neuroblastoma response. The response rate to the induction phase of the regimen and a corresponding 95% confidence interval will be calculated for all strata combined.
Time Frame: 12 weeks after participant received the first dose
Population: Ineligible patients were excluded from analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Eligible Patients: All eligible Stage 2/3, Stage 4a, and Stage 4b patients
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 57
percentage of participants | 68 [56 to 79]

3. Secondary Outcome: Percentage of Participants With Adverse Events as Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Grade 3 and higher toxicities will be descriptively summarized.
Time Frame: Up to 30 days after completion of study treatment
Population: Three ineligible patients were excluded from this analysis. Two patients who did not receive therapy were also excluded from this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Stage 2/3 Patients | Stage 4a Patients | Stage 4b Patients
Number analyzed (Participants) | 18 | 18 | 19
percentage of participants
  Abdominal pain | 0 | 5.6 | 0
  Acute kidney injury | 0 | 5.6 | 0
  Alanine aminotransferase increased | 0 | 16.7 | 5.3
  Anemia | 0 | 0 | 5.3
  Anorexia | 11.1 | 33.3 | 15.8
  Apnea | 0 | 0 | 5.3
  Aspartate aminotransferase increased | 0 | 11.1 | 5.3
  Catheter related infection | 11.1 | 0 | 0
  Dehydration | 0 | 11.1 | 10.5
  Depressed level of consciousness | 0 | 0 | 5.3
  Diarrhea | 5.6 | 16.7 | 0
  Encephalopathy | 0 | 0 | 5.3
  Enterocolitis | 0 | 5.6 | 0
  Enterocolitis infectious | 5.6 | 11.1 | 5.3
  Esophagitis | 0 | 5.6 | 0
  Febrile neutropenia | 55.6 | 55.6 | 36.8
  Fever | 11.1 | 0 | 5.3
  GGT increased | 0 | 5.6 | 0
  Gastric hemorrhage | 0 | 5.6 | 0
  Hearing impaired | 11.1 | 5.6 | 5.3
  Hypermagnesemia | 5.6 | 0 | 0
  Hypertension | 0 | 5.6 | 0
  Hypoalbuminemia | 0 | 0 | 5.3
  Hypocalcemia | 5.6 | 5.6 | 10.5
  Hypoglycemia | 0 | 0 | 5.3
  Hypokalemia | 27.8 | 16.7 | 21.1
  Hypomagnesemia | 5.6 | 5.6 | 10.5
  Hyponatremia | 11.1 | 0 | 15.8
  Hypophosphatemia | 22.2 | 0 | 10.5
  Hypotension | 0 | 11.1 | 0
  Hypoxia | 0 | 2.6 | 0
  Infections and infestations - Other, specify | 27.8 | 33.3 | 21.1
  Lower gastrointestinal hemorrhage | 0 | 5.6 | 0
  Lung infection | 16.7 | 0 | 0
  Lymphocyte count decreased | 0 | 0 | 5.3
  Mucositis oral | 5.6 | 27.8 | 5.3
  Nausea | 16.7 | 11.1 | 5.3
  Nervous system disorders - Other, specify | 0 | 0 | 10.5
  Neutrophil count decreased | 5.6 | 0 | 5.3
  Oral pain | 0 | 5.6 | 0
  Pain | 0 | 5.6 | 0
  Peripheral motor neuropathy | 5.6 | 0 | 0
  Pharyngeal mucositis | 0 | 5.6 | 0
  Platelet count decreased | 5.6 | 0 | 5.3
  Pneumonitis | 5.6 | 0 | 0
  Rectal pain | 0 | 5.6 | 0
  Seizure | 0 | 0 | 5.3
  Sepsis | 0 | 11.1 | 0
  Sinus tachycardia | 0 | 5.6 | 0
  Sinusitis | 11.1 | 0 | 0
  Skin infection | 0 | 5.6 | 5.3
  Upper respiratory infection | 11.1 | 5.6 | 0
  Vomiting | 11.1 | 22.2 | 5.3
  White blood cell decreased | 5.6 | 0 | 5.3

ADVERSE EVENTS:
Time Frame: Up to 30 days after completion of study treatment.
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution, via expedited reporting (NCI AdEERs / CAeRs). The "AE Other" table reflects all CTCAEs collected excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Stage 2/3 Patients | Stage 4a Patients | Stage 4b Patients
All-Cause Mortality (participants affected / at risk) | 2/18 | 5/18 | 15/19
Serious Adverse Events (participants affected / at risk) | 1/18 | 2/18 | 0/19
Other Adverse Events (participants affected / at risk) | 13/18 | 12/18 | 10/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 2/3 Patients (N=18) | Stage 4a Patients (N=18) | Stage 4b Patients (N=19)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 2/3 Patients (N=18) | Stage 4a Patients (N=18) | Stage 4b Patients (N=19)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 3 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 6 | 3
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1
Catheter related infection (Infections and infestations) | 2 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 3 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 2 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 9 | 7
Fever (General disorders) | 2 | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
GGT increased (Investigations) | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 2 | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 5 | 3 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 0 | 2
Hypotension (Vascular disorders) | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 5 | 6 | 4
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Lung infection (Infections and infestations) | 3 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 5 | 1
Nausea (Gastrointestinal disorders) | 3 | 2 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 1
Upper respiratory infection (Infections and infestations) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 1
White blood cell decreased (Investigations) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT00554788/Prot_SAP_000.pdf